CLINICAL TRIAL: NCT04997681
Title: SYNchronizing Exercises, Remedies in Gait and Cognition at Home: Feasibility of a Home-based Double-blind Randomized Controlled Trial to Improve Gait and Cognition in Individuals at Risk for Dementia
Brief Title: SYNchronizing Exercises, Remedies in Gait and Cognition at Home (SYNERGIC@Home)
Acronym: SYNERGIC@Hom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Horizon Health Network (Other); Réseau de Santé Vitalité Health Network (Other); Universite de Moncton (Other); Western University, Canada (Other)
Responsible Party: Principal Investigator, Chris A. McGibbon, PhD, Professor, University of New Brunswick
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: SYNH001
Record Dates: First submitted 2021-06-01; First posted 2021-08-10 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Exercise; Cognitive training; Intervention preference; Elderly; Gait; Dementia; Home-based intervention; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Dementia | interventions — Resistance Training; Cognitive Training

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise Intervention Training and Cognitive Intervention Training (Experimental): Combined Aerobic Exercise and Resistance Training (AE + RT) + Cognitive Training (NeuropeakTM)
  Interventions: Behavioral: Combined Aerobic Exercise and Resistance Training (AE + RT); Behavioral: Cognitive Training (NeuropeakTM)
- Exercise Intervention Training and Control Cognitive Training (Active Comparator): Combined Aerobic Exercise and Resistance Training (AE + RT) + Control Cognitive Training of Website Searching and Video Watching (WS+V)
  Interventions: Behavioral: Combined Aerobic Exercise and Resistance Training (AE + RT); Behavioral: Control Cognitive Training of Website Searching and Video Watching (WS+V)
- Control Exercise Training and Cognitive Intervention Training (Active Comparator): Control Balance and Toning Exercise Training (BAT) + Cognitive Training (NeuropeakTM)
  Interventions: Behavioral: Cognitive Training (NeuropeakTM); Behavioral: Control Balance and Toning Exercise Training (BAT)
- Control Exercise Training and Control Cognitive Training (Placebo Comparator): Control Balance and Toning Exercise Training (BAT) + Control Cognitive Training of Website Searching and Video Watching (WS+V)
  Interventions: Behavioral: Control Cognitive Training of Website Searching and Video Watching (WS+V); Behavioral: Control Balance and Toning Exercise Training (BAT)

INTERVENTIONS:
Behavioral: Combined Aerobic Exercise and Resistance Training (AE + RT) — AE + RT will be conducted via a video-conferencing platform under the direct supervision and coaching of a certified exercise physiologist with certification from the Canadian Society for Exercise Physiology (CSEP; or equivalent certification). These certified trainers will administer the exercise interventions in a one trainer to one participant ratio. AE + RT includes a set of warm up exercises, which will be completed in approximately 5 minutes, followed by a break. Next, 6 strength training exercises (that progressively increase in resistance intensity over time) will be completed followed by a break. Aerobic exercises that safely increase the participant's heart rate will follow for 30 minutes followed by a break and a set of cool down exercises for 5 minutes. In total the AE + RT exercise session is approximately 65 minutes.
  Arms: Exercise Intervention Training and Cognitive Intervention Training; Exercise Intervention Training and Control Cognitive Training
Behavioral: Cognitive Training (NeuropeakTM) — NeuropeakTM is a program which will be completed by participants remotely using a tablet or computer. It consists of cognitive training including dual-task training that requires participants to maintain and prepare for many response alternatives (working memory) and to share attention between two concurrent tasks (divided attention). Difficulty of cognitive training is tailored to their individual functioning level. During each session, participants perform one of two different visuo-motor tasks, which include sets of visual stimuli (e.g., letters, numbers, animals, vehicles, fruits, celestial bodies) and respective hand-button correspondences (i.e., keys that are to be tapped on either the right or the left side of the screen). Participants are instructed to perform these tasks as fast as possible, while maintaining accuracy. Training also includes online feedback and a histogram of daily performance to encourage improvement. NeuropeakTM takes approximately 30 minutes to complete.
  Arms: Control Exercise Training and Cognitive Intervention Training; Exercise Intervention Training and Cognitive Intervention Training
Behavioral: Control Cognitive Training of Website Searching and Video Watching (WS+V) — During the WS + V task, participants alternate between 2 different tasks (touristic searching using internet and video watching). For the touristic searching using internet, participants are required to find 3 hotels, 3 touristic places, and 3 restaurants of their own preference in a city assigned by the instructor (a new city will be selected each session). They will also need to include the respective addresses of those places on their log sheet. For the video watching task, participants watch a National Geographic video on YouTube selected by the instructor with a different video selected for each session. They will watch the video for 20 minutes and during the remaining 5 minutes they will answer the following questions on their log sheet: 1) What is the video about? 2) What is the most important information in your opinion? 3) Create a question based on the video and answer your own question. WS + V sessions take approximately 30 minutes to complete.
  Arms: Control Exercise Training and Control Cognitive Training; Exercise Intervention Training and Control Cognitive Training
Behavioral: Control Balance and Toning Exercise Training (BAT) — BAT exercises will be conducted via a video-conferencing platform under the direct supervision and coaching of a certified exercise physiologist with certification from the Canadian Society for Exercise Physiology (CSEP; or equivalent certification). These certified trainers will administer the exercise interventions in a one trainer to one participant ratio. BAT includes a set of warm up exercises, which will be completed in approximately 5 minutes, followed by a break. Next, 6 balance and toning exercises will be completed followed by a break. Stretching exercises will follow for 30 minutes followed by a break and a set of cool down exercises for 5 minutes. In total the BAT exercise session is approximately 65 minutes.
  Arms: Control Exercise Training and Cognitive Intervention Training; Control Exercise Training and Control Cognitive Training

SUMMARY:
Background: Prevention of Alzheimer's Disease and Related Dementias (ADRDs) may be possible for persons with subjective (SCI) or mild cognitive impairment (MCI), or normal cognition and risk factors. Physical exercise and cognitive training have been shown to enhance cognitive function and mobility in MCI when delivered in a research facility. The feasibility of delivering interventions in the home of older adults at risk for developing ADRDs is not known. What preferences the participants have for these interventions are also unknown. The primary goals are: 1) assess feasibility of a home-based delivery of exercise and cognitive interventions 2) evaluate the relationship between participants' intervention preferences and adherence. Secondary objectives focus on cognition, frailty, mobility, sleep, diet and mental health.

Methods and analysis: SYNERGIC@Home is a randomized control trial (using a 2 x 2 factorial design) with a 16-week home-based intervention program of physical exercises with cognitive training. Sixty-four participants will be randomized in blocks of four: 1) combined exercise (aerobic and resistance) + cognitive training (NEUROPEAK™); 2) combined exercise + control cognitive training (web searching); 3) control exercise (balance and toning) + cognitive training; and 4) control exercise + control cognitive training. It will be implemented virtually through video conferencing. Baseline, 4- and 10-month post-intervention will include measures of cognition, frailty, mobility, sleep, diet, and psychological health. Feasibility outcomes include recruitment and retention. Preference will be used to determine the relationship between preference adherence. Secondary outcomes will evaluate the effect of the interventions on cognitive, mobility, and general well-being.

DETAILED DESCRIPTION:
BACKGROUND: Nearly half a million Canadians live with Alzheimer's Disease and Related Dementias (ADRDs), and approximately one third of those cases could have been prevented with early intervention. Physical exercise and cognitive training are emerging interventions that have the potential to enhance cognitive function and mobility in older adults at risk for developing dementia. The SYNERGIC trial (SYNchronizing Exercises, Remedies in GaIt and Cognition), a large multi-site randomized control trial, showed promising preliminary data that individuals in an active exercise intervention combining aerobic exercise with progressive resistance training (AE+RT) and in a cognitive training program (NEUROPEAKTM) had better cognitive outcomes than a balance and toning control (BAT) intervention paired with a control cognitive intervention consisting of website searching and watching a simple video (WS+V). While these interventions were provided face to face in a research facility, little is known about the feasibility of delivering these multi-domain interventions at home in older adults at risk for developing ADRDs. Thus, the primary goal of the present trial-the SYNERGIC@Home trial-is to establish the feasibility of delivering a combined multimodal exercise and cognitive training intervention program for 16 weeks to 64 older adults at home using video-conferencing.

HYPOTHESIS: Based on the success of the SYNERGIC trial, we expect that SYNERGIC@Home will follow suit and yield high recruitment, retention, and adherence rates-particularly in light of the fact that SYNERGIC@Home eliminates any of the natural inconveniences of in person testing.

METHODS: SYNERGIC@Home is a randomized control trial (RCT) with a 16-week home-based intervention program of combined physical exercises with cognitive training. Sixty-four participants will be randomized to one of the following four arms: 1) combined exercise (AE+RT) + cognitive training (NEUROPEAKTM); 2) combined exercise (AE+RT) + control cognitive training (WS+V); 3) Control exercise (BAT) + cognitive training (NEUROPEAKTM) ; and 4) Control exercise (BAT) + control cognitive training (WS+V). SYNERGIC@Home will be implemented entirely virtually through video and phone conferencing. Baseline, immediate post-intervention follow-up, and 6-month post-intervention follow-up assessments will include measures of cognition, frailty, mobility, sleep, diet, and psychological health. For primary feasibility objectives, we will obtain measures of recruitment and retention rates. For primary analytic objectives, we will examine the distribution of preference ratings and determine if there is a relationship between preference for a given intervention and subsequent adherence. A series of secondary analytic outcomes examining the potential effect of the individual and combined interventions on cognitive, mobility, and general well-being will be measured at both baseline and follow-up. If we find a relatively equal split in sex our sample, we will conduct gender-based analyses as additional, exploratory research.

EXPECTED RESULTS AND DISCUSSION: The SYNERGIC@Home trial will establish the feasibility of a combined multimodal intervention program delivered at home in older adults. Similarly, it will estimate the frequency and strength of participant preference for different interventions and delineate the relationship between intervention preference and subsequent adherence. It will also build capacity for and pilot the delivery of multi-domain interventions using an entirely home-based protocol with individuals at risk for ADRDs. The SYNERGIC@Home trial will inform future larger scale studies on the feasibility and success of implementing home-based interventions for individuals at risk for ADRDs. Insights gained from this feasibility trial will be instrumental in developing various other at home, remote, and virtual intervention programs for community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 to 90 years old.
* Has a Family Physician
* Has internet access (and have regular access to email), and the technology ability (able to send and receive emails).
* Resides in their own home/apartment in the community.
* Has access to a home computer and/or a tablet computer device.
* Self-reported levels of proficiency in English and/or French for speaking and understanding spoken and written language.
* Able to comply with scheduled home-based assessments, interventions, and other trial procedures.
* Able to ambulate at least 10 m independently with or without a walking aid.
* Being at risk of developing dementia:

  1. Mild Cognitive Impairment (MCI) Group. Diagnosis of Mild Cognitive Impairment, in accordance with the criteria used in the Comprehensive Assessment of Neurodegeneration and Dementia (COMPASS-ND) study2 (Table 1).
  2. Subjective Cognitive Impairment (SCI) Group. Diagnosis of Subjective Cognitive Impairment, in accordance with the COMPASS-ND study2 definition (Table 1).
  3. Cognitively Intact with Risk Factors Group. Cognitively Intact based on COMPASS ND study2 definition (Table 1)) AND have a history of two or more risk factors for dementia, defined as the following (Table 1):

     * Obesity: Defined as a Body Mass Index (BMI) > 30 kg/m2 (as derived from the National Institute of Health BMI calculator52)
     * Hypertension: Defined as a documented Systolic Blood Pressure > 140 mm Hg, OR a physician's diagnosis of hypertension, OR presence of physician prescribed medical treatment for hypertension, OR other approaches to treatment for hypertension (i.e., diet or exercise).
     * Diabetes: Defined as a physician's diagnosis of diabetes, OR presence of physician prescribed medical treatment for diabetes, OR other approaches to treatment for diabetes (i.e., diet or exercise).
     * Cardiovascular disease: Defined as a physician's diagnosis of angina, myocardial infarction, coronary revascularization or other arterial revascularization, stroke, transient ischemic attack and/or peripheral vascular disease.
     * Physical inactivity: Defined as inactive, whereby active is defined as engaging in a minimum of 20-30 minutes of physical activity causing sweating and breathlessness, at least two times per week.
     * First-degree family history of dementia: Defined as a physician's diagnosis of dementia in a first-degree relative, including a parent, sibling, or child.
     * Dyslipidemia: Defined as a documented total cholesterol > 6.5 mmol/L, OR a physician's diagnosis of hypercholesterolemia, OR presence of physician prescribed medical treatment for hypercholesterolemia, OR other approaches to treatment (e.g. diet, exercise).
     * Poor sleep: Defined as a score of 6 or higher on the PSQI-18 (higher scores indicate poorer sleep).
     * Poor diet: Defined as a score of 7 or less on the MDA-14.
* Must be medically able to participate in the study's exercise training program, as determined using the Get Active Questionnaire (a screening tool developed by the Canadian Society for Exercise Physiology53), coupled with evaluation by a certified exercise physiologist and/or the study physician for clearance to participate in combined exercise training program.
* Preserved activities of daily living operationalized as a score of > 14/23 on the Lawton-Brody Instrumental Activities of Daily Living (IADL) scale3 and confirmed by clinician's interviews.

Exclusion Criteria:

* A diagnosis of dementia
* Participants living in Nursing Homes or Adult Residential Facilities (Special Care Homes) will be excluded.
* Serious underlying disease, which, in the opinion of the study physician excludes engagement in interventions or may interfere with the participant's ability to participate fully in the study.
* Has had surgery within the last two months or has planned surgery in the coming 12 months that, deemed by the study physician, could interfere with the participant's vision, hearing, mobility or any other ability to participate in the study.
* Has a history of intracranial surgery.
* Regular Benzodiazepine use by a participant that the study physician determines to be significant enough to interfere with the participants ability to participate in the assessments and interventions in the study will be excluded.
* Presence of major depression, schizophrenia, severe anxiety or drug/alcohol abuse, or other medical illness that would prohibit them from safely participating in the study or may cause harm to the participant.
* Current Parkinsonism or any neurological disorder with residual motor deficits (e.g. stroke with motor deficit), active musculoskeletal disorders (e.g. severe osteoarthritis of lower limbs), or history of knee/hip replacement affecting gait performance during the baseline assessment.
* Severe visual and/or auditory impairment, which, according to the vision and hearing assessment, precludes the participant from engaging in the trial.
* Intention to enroll in other clinical trials during the same time period.
* Active participation in an organized and planned exercise program involving aerobic exercise and/or resistance training regimen in the previous 6 months.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Intervention Adherence | Post-intervention at 4 months
  Defined as the mean percent of all Intervention sessions attended of the 48 planned sessions per participant.
Intervention Preference | Baseline
  The primary analytic goal of SYNERGIC@Home is to assess the relationship between participants' adherence to the interventions and their affinity for each intervention going into the trial. All participants will be given the Intervention Preference Questionnaire (IPQ) prior to implementation of the intervention

SECONDARY OUTCOMES:
Recruitment Rate | Through study completion, an average of 10 months
  Defined as the total percent of enrolled participants relative to number of people screened for eligibility.
Retention Rate | Through study completion, an average of 10 months
  Defined as the total percent of enrolled participants who continue throughout the trial and participate in outcomes assessments as follows:
  * Enrollment retention: of those enrolled participants, the % who complete immediate 4-month post intervention assessment, and;
  * Follow-up retention: of those who complete the immediate 4-month post intervention follow-up assessment, the % of participants who complete the 6-month post-intervention follow-up assessment at 10-months.
Assessment Tolerability | Baseline
  Defined as total percent of participants not voluntarily dropping out during baseline or between baseline assessment and prior to allocation to intervention group.
Trial Experience | 10 months follow-up
  Trial experience is defined as participants' qualitative responses to semi-structured open-ended questions aimed at providing insights on their overall trial experience within the context of the Kirkland evaluation framework.
Adverse Events | Monitored from start of study until end of study
  Frequency cross-tabulation of AE severity versus AE relation to trial.
Height | Baseline
  This measurement will be done at home and self-reported.
Data Loss | Through study completion, an average of 10 months
  Defined as data lost due to technical failures, personnel errors or participant non-compliance
Weight | Baseline
  This measurement will done at home and self-reported.
Sex | Baseline
  This measurement will be self-reported.
Age | Baseline
  This measurement will be self-reported.
Change in Hip Circumference | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This measurement will be done at home and self-reported.
Change in Neck Circumference | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This measurement will be done at home and self-reported.
Change in waist circumference | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This measurement will be done at home and self-reported.
Change in blood pressure | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Measured with a provided blood pressure cuff. Reported systolic/diastolic.
Change in heart rate | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Measured with a provided blood pressure cuff. Reported in beats/minute.
Change in Medications | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This measurement will be self-reported.
Chronic Diseases | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This measurement will be self-reported and will be monitored throughout the trial
Change in fall history | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Falls will be recorded throughout the trial, in which participants will be provided with a falls calendars, on which they will record any falls that have occurred, and the research team will collect them monthly.
Change in Health Status and Self-Perception | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on their self-perception of their health status
Change in Constant Fatigue | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on fatigue.
Change in Falls and Balance | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on falls and balance
Change in Vision | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on their vision
Change in Hearing | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on their hearing
Change in Nutrition | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on their nutrition.
Change in Sleep | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on their sleep.
Change in Mayo Fluctuation Scale | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will answer questions on how they feel during a day. Scores range between 0 and 4 with higher scores meaning a worse outcome.
Change in Telephone Cognitive Screen (TCogS) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  is a widely used tool that measures cognitive function in older individuals. The telephone version of the CogS has been standardized and will be administered via video conferencing. It consists of a 26-point assessment that measures orientation, registration, attention and calculation, recall, and language
Change in Clinical Dementia Rating Scale (CDR) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The CDR is a validated 5-point composite scale used in longitudinal Alzheimer's Disease (AD) research to characterize cognitive and global function performance applicable to AD and related dementias.61 Information is obtained through a semi-structured interview of the patient and a reliable informant or collateral source (e.g. family member).
Change in remote version of the Montreal Cognitive Assessment (MoCA) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The Full MoCA via Audio-Visual Conference consists of a 30-point test assessing the following items: short term memory recall, visuospatial abilities, executive functioning, phonemic fluency, verbal abstraction, attention, concentration, working memory, language, and orientation.
Change in Lawton-Brody Instrumental Activities of Daily Living (IADL) scale | Baseline, post-intervention at 4 months, and follow-up at 10 months
  measures participant's ability to engage in instrumental activities of daily living via questionnaire assessing activities such as preparing meals and managing personal finances
Change in ADAS-Cog Immediate Word Recall | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants are presented with 10 high imagery words and are given three trials to learn and recall them.
Change in ADAS-Cog Delayed Word Recall | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants are asked to recall the 10 high imagery words presented during the immediate word recall task after a delay of approximately 5 to 10 minutes.
Change in ADAS-Cog Orientation | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants are asked 8 questions pertaining to their identity, the place, and the time.
Change in Cognitive Functional Composite 2 (CFC-2) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The CFC-2 is a collective of different test which consists of the ADAS-Cog Immediate Word Recall, ADAS-Cog Delayed Word Recall, ADAS-Cog Orientation, Clinical Dementia Rating Sum of Boxes (CDR-SB) Cognitive portion, and the Functional Activities Questionnaire.
Functional Activities Questionnaire | Baseline, post-intervention at 4 months, and follow-up at 10 months
  It measures participant's ability to engage in instrumental activities of daily living via questionnaire assessing activities such as preparing meals and managing personal finances
Change in Oral Trail Making Test (TMT) A | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The Oral Trail Making Test (TMT) A & B is a two-part test that assesses attention speed, and mental flexibility and has been widely used in clinical settings for assessing deficits in attention and executive functioning.
Change in Oral Trail Making Test (TMT) B | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The Oral Trail Making Test (TMT) A & B is a two-part test that assesses attention speed, and mental flexibility and has been widely used in clinical settings for assessing deficits in attention and executive functioning.
Change in 15-item Boston Naming Test (BNT) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The Boston Naming Test (BNT) assesses visual confrontational naming and asks participants to name simple line drawings of objects.
Change in Logical Memory I | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Logical Memory I & II (Story A) from the Wechsler memory scale assesses memory and free recall. Scores range between 0 and 25 with higher scores meaning a better outcome.
Change in Logical Memory II | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Logical Memory I & II (Story A) from the Wechsler memory scale assesses memory and free recall. Scores range between 0 and 25 with higher scores meaning a better outcome.
Change in ADAS-Cog Word Recognition | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants are presented with a list of 12 words and are then asked to identify the words among a list of distractor words.
Change in The Delis-Kaplan Executive Function System (DKEFS) phonemic fluency test | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The Delis-Kaplan Executive Function System (DKEFS) phonemic fluency test measures phonemic verbal fluency.
Change in The Delis-Kaplan Executive Function System (DKEFS) semantic fluency test | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The Delis-Kaplan Executive Function System (DKEFS) semantic fluency test measures speed and flexibility of verbal thought.
Change in Digit Span Backward Test | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The digit span test is an auditory attention task, in which participants are asked to recall a series of numbers forward and backward.
Change in Oral version of the Digit Symbol Modalities Test | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This is a timed task that gives participants 120 seconds to orally match geometric figures with specific numbers according to a defined key (specifying which symbols are assigned to which numbers) that is provided at the top of the stimulus page.
Change in 18-item Pittsburgh Sleep Quality Index (PSQI-18) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This is a 18-item questionnaire to help evaluate a participants sleep quality
Change in Work and Sleep Diary (WSD) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A self reported work and sleep diary to track activity and sleep during the assessments.
Change in 14-item Mediterranean Diet Assessment (MDA-14) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A 14-item questionnaire to help evaluate a participants diet.
Change in Eating Pattern Self-Assessment | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The Eating Pattern Self-Assessment is a tool used for participants to provide a self-report on their eating patterns.
Change in Questionnaire for Vitamin D intake | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A questionnaire to determine a participant's intake of Vitamin D.
Change in Physical Activity Scale for the Elderly (PASE) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A questionnaire to assess a participants activity level. Scores range from 0 to 400+ with higher scores meaning a better outcome.
Change in Life Space Questionnaire (LSQ) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A questionnaire to assess a participant's mobility ability.
Change in Clinical Frailty Scale (CFS) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  This assessment will be performed by the Clinical Research Coordinator/nurse using the 9 point CFS instrument. This will allow for a determination of the clinical frailty of the participants. Scores range between 1 and 9 with higher scores meaning a worse outcome.
Change in Short Form quality of life questionnaire (SF-36) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A 36-item questionnaire that evaluates different aspects of quality of life.
COVID-19 Questionnaire | Baseline
  A questionnaire that assesses a participants experience with the current COVID-19 pandemic. Scores range from 10-40 when self reported or 8-33 when reported by a study partner.
Change in Generalized Anxiety Disorder 7 (GAD 7) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A questionnaire to establish a participant's experience with anxiety
Change in Geriatric Depression Scale (GDS-30) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  A questionnaire to establish a participant's experience with depression
Short Test of Functional Health Literacy in Adults (STOFHLA) | Baseline
  Health Literacy will be assessed using the abbreviated version of the Test of Functional Health Literacy in Adults (TOFHLA).The short version, STOFHLA, consists of 2 prose passages and 4 numeracy items.
Change in Functional Assessment of Currently Employed Technology Scale (FACETS) | Baseline, post-intervention at 4 months, and follow-up at 10 months
  The FACETS is a 10-item questionnaire with possible responses falling on a Likert-type scale, and higher scores indicating more frequent use of technology domains.
Change in seated dual task | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will be asked to name as many animals as they are able to, count backwards by 1's, and count backwards by 7's while seated.
Change in single-task gait | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Their gait velocity will be measured 3 times. Gait variability of spatial and temporal gait variables (stride time, stride length, double support time and step width) will be measured and the coefficient of variation calculated (CV = (standard deviation / mean) x 100).
Change in dual-task gait | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will perform three walks, once each under the following dual-task conditions: walking while naming animals, counting backwards from 100 by 1's, and counting backwards from 100 by 7's.
Change in Sit to Stand Test (STST) performance | Baseline, post-intervention at 4 months, and follow-up at 10 months
  Participants will be asked to sit and stand, from a chair, repetitively for 60 seconds.
Biomarkers of Alzhiemer's Disease and Related Diseases | Post intervention, at 8 months
  A saliva sample will be taken to get a Polygenic Hazard Score is derived from a panel of 31 single nucleotide polymorphisms. The genetic content known as DNA, or deoxyribonucleic acid, will be analyzed in order to learn about genetic information that may increase a person's risk for developing dementia. This test is part of the overall outcome measure and is not a diagnostic test. Study participants will not receive results of this test. This test is not currently a standard of normal clinical care and is still under research to determine its utility in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Chris McGibbon, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- The University of New Brunswick, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be stored on a secure server called LORIS (Longitudinal Online Research and Imaging System) at the McGill Centre for Integrative Neuroscience, McGill University, Montreal, Quebec.
Supporting Information: Study Protocol
Time Frame: 12 months after the principal paper answering primary research questions are published.
Access Criteria: Qualified persons may request access via email to the Canadian Consortium for Neurodegeneration and Aging [ccna.admin@ladydavis.ca].

REFERENCES:
- [Derived] Omar H, Yetman L, Tranchant CC, Gallibois M, Hache JC, Faig K, Handrigan G, McGibbon C, Jarrett P. "It's About Connections": A Grounded Theory of Older Adults' Engagement in Remotely Delivered Home-Based Physical and Cognitive Exercise Interventions Aiming to Reduce the Risk of Dementia. J Patient Exp. 2025 Oct 30;12:23743735251392324. doi: 10.1177/23743735251392324. eCollection 2025. PMID 41180905
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] McGibbon C, Jarrett P, Handrigan G, Bouchard D, Tranchant CC, Sexton AM, Yetman L, Robinson B, Crapoulet S, Chamard-Witkowski L, Liu-Ambrose T, Middleton LE, Almeida QJ, Bherer L, Lim A, Speechley M, Kamkar N, Montero Odasso M; Canadian Consortium on Neurodegeneration in Aging (CCNA), CAN-THUMBS UP Group. Protocol for SYNchronising Exercises, Remedies in GaIt and Cognition at Home (SYNERGIC@Home): feasibility of a home-based double-blind randomised controlled trial to improve gait and cognition in individuals at risk for dementia. BMJ Open. 2022 Mar 31;12(3):e059988. doi: 10.1136/bmjopen-2021-059988. PMID 35361653